CLINICAL TRIAL: NCT06316856
Title: CD5 Chimeric Antigen Receptors (CAR) T Cells in Subjects With Relapsed or Refractory T-Cell Malignancies: a Multi-center, Open-label, Non-randomized, Phase 1/2 Clinical Trial
Brief Title: CD5 Chimeric Antigen Receptor (CAR) T Cells in Subjects With Relapsed or Refractory T-cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: The General Hospital of Western Theater Command (Other); Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai (Other); Shanghai Liquan Hospital (Other); Central People's Hospital of Zhanjiang (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2024-002
Record Dates: First submitted 2024-03-10; First posted 2024-03-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: T-Cell Acute Lymphocytic Leukemia; Acute Lymphoblastic Leukemia, in Relapse; Refractory Acute Lymphoblastic Leukemia; T-cell Malignancies
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autologous CD5 CAR T-cells (Experimental): After a lymphodepleting regimen, the patients will receive autologous CD5 CAR T-cell infusion.
  Interventions: Drug: Autologous CD5 CAR T-cells
- Prior stem-cell transplantation (SCT) donor-derived CD5 CAR T-cells (Experimental): After a lymphodepleting regimen, the patients will receive prior SCT donor-derived CD5 CAR T-cell infusion.
  Interventions: Drug: Previous stem-cell transplantation (SCT) donor-derived CD5 CAR T-cells
- Newly matched donor-derived CD5 CAR T-cells (Experimental): After a lymphodepleting regimen, the patients will receive newly matched donor-derived CD5 CAR T-cell infusion.
  Interventions: Drug: Newly matched donor-derived CD5 CAR T-cells

INTERVENTIONS:
Drug: Autologous CD5 CAR T-cells — Peripheral blood mononuclear cells for the production of CD5 CAR T-cells from patients.
  Arms: Autologous CD5 CAR T-cells
Drug: Previous stem-cell transplantation (SCT) donor-derived CD5 CAR T-cells — Peripheral blood mononuclear cells for the production of CD5 CAR T cells are collected from previous SCT donors.
  Arms: Prior stem-cell transplantation (SCT) donor-derived CD5 CAR T-cells
Drug: Newly matched donor-derived CD5 CAR T-cells — Peripheral blood mononuclear cells for the production of CD5 CAR T cells are collected from newly matched donors.
  Arms: Newly matched donor-derived CD5 CAR T-cells

SUMMARY:
This is a multi-center, open-label, non-randomized, phase 1/2 study of anti-CD5 CAR-T cell therapy in patients with CD5+ relapsed or refractory T-cell malignancies. A bayesian optimal interval (BOIN) 12 design will be used to explore the optimal biological dose (OBD) from starting dose level 1: 1×10^6 (±20%) to dose level 2: 2×10^6 (±20%) in three cohorts (autologous, previous-transplant-donor or newly matched donor-derived CD5 CAR T cells). If the manufactured cells are not sufficient to meet the preassigned standard dose criteria, patients will be given infusion at a low dose level of 5×10^5 (±20%) /kg. The primary objective is to evaluate the safety and tolerability of CD5 CAR T cell therapy in subjects, determine the OBD and recommend phase 2 dose (RP2D) in phase 1, and evaluate the efficacy of CD5 CAR T cell therapy in phase 2. The primary endpoint is the type and incidence of dose-limiting toxicity (DLT) within 28 days, and the incidence and severity of adverse events (AEs) within 30 days after CD5 CAR T-cell infusion in phase 1, the best overall response (BOR) at 3 months (± 1 week) after CD5 CAR T-cell infusion in phase 2. A total number of 54 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Only patients who meet all the following criteria can be included:

1. Candidates with relapse or refractory CD5+ T-cell malignancies, who have progressed after treatment with all standard therapies or been intolerant of standard care, have limited prognosis with currently available therapies and have no available curative treatment options (such as stem-cell transplantation (SCT) or chemotherapy);
2. For subjects who received autologous CD5 CAR T cells, the tumor burden in peripheral blood is less than 20%, and suspending anti-neoplastic treatment for more than 2 weeks;
3. Aged 1-70 years;
4. No severe allergy;
5. Eastern Cooperative Oncology Group (ECOG) performance status 1 score 0 to 2;
6. Patients are expected to live for at least 60 days;
7. CD5+ on blasts in bone marrow (BM) or cerebrospinal fluid (CSF) and tumor tissues by flow cytometry and immunohistochemistry, respectively. (Positive rate >80% by flow cytometry with less than one log difference in mean fluorescence intensity from normal T cells, or positive rate >30% positive by immunohistochemistry);
8. Provide a signed informed consent before any screening procedure. Subjects who voluntarily participate in the study should have the ability to understand and sign the informed consent form and be willing to follow the study visit schedule and relevant study procedure, as specified in the protocol. Candidates aged 19-70 years need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form. Children candidates of 8-18 years old need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form and their legal guardian or patient advocate has also need to sign the treatment consent form and voluntary consent form, respectively. Children candidates of 1-7 can be recruited after the legal guardian or patient advocate has signed the treatment consent form and voluntary consent form;
9. Have available allogeneic hematopoietic stem cell transplantation donor for the subject who received newly matched donor-derived CD5 CAR T cells, and is willing to perform SCT when CR is achieved.

Exclusion Criteria:

Patients with at least one of the following conditions are excluded:

1. Impaired consciousness or intracranial hypertension;
2. Symptomatic congestive heart failure or severe cardiac arrhythmia;
3. Manifestations of severe respiratory system failure;
4. Co-existence with other malignancies;
5. Disseminated intravascular coagulation;
6. Serum creatinine and/or blood urea nitrogen (BUN) ≥ 1.5-fold upper limit;
7. Sepsis or other uncontrollable infections;
8. Uncontrollable diabetes;
9. Serious mental illness;
10. Apparent and active intracranial lesions on cranial magnetic resonance imaging (MRI);
11. Underwent organ transplantation, excepting SCT;
12. Pregnant females;
13. Positive test for infectious hepatitis, acquired immune deficiency syndrome (AIDS) or syphilis;
14. Post-CAR SCT is not feasible in patients who plan to receive newly matched donor-derived CD5 CAR T cells;
15. Inability to collect peripheral blood mononuclear cells (PBMC) or no frozen PBMC available for CAR T cell manufacturing.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1-The incidence and type of dose-limiting toxicity (DLT) | 28 days after CD5 CAR T cell infusion
  The number of patients experiencing dose-limiting toxicity (DLT) will be evaluated and the type of DLT will be recorded.
Phase 1-The incidence and severity of adverse events (AEs) | 30 days after CD5 CAR T cell infusion
  The number of patients experiencing adverse events (AEs) and the severity of AEs will be evaluated.
Phase 2-Antitumor effect | 3 months (± 1 week) after CD5 CAR T infusion
  Assessment of best overall response (BOR) rate. BOR rate is the percentage of patients with the best overall response in complete response (CR), complete response with incomplete hematological recovery (CRi) or partial response (PR) based on the National Comprehensive Cancer Network (NCCN) Guidelines Version 3.2023 of Acute Lymphoblastic Leukemia.

SECONDARY OUTCOMES:
Phase 1-Objective response rate (ORR) | 30 days after CD5 CAR T cell infusion
  Objective response rate (ORR) is the percentage of subjects who have achieved CR, CRi or PR based on the National Comprehensive Cancer Network (NCCN) Guidelines Version 3.2023 of Acute Lymphoblastic Leukemia.
Phase 1-Pharmacokinetics of CD5 CAR T cells | Up to 2 years after CD5 CAR T cell infusion
  The proliferation and survival of CAR T cells will be measured by flow cytometry and quantitative polymerase chain reaction (qPCR).
Phase 1-The incidence and severity of adverse events (AEs). | From 30 days to 2 years after CD5 CAR T cell infusion
  The number of patients experiencing adverse events (AEs) and the severity of AEs will be evaluated.
Phase 1-Best overall response (BOR) rate. | 3 months (± 1 week) after CD5 CAR T cell infusion
  BOR rate is the percentage of patients with the best overall response in CR, CRi or PR based on the National Comprehensive Cancer Network (NCCN) Guidelines Version 3.2023 of Acute Lymphoblastic Leukemia.
Phase 2-Objective response rate (ORR) | 1 months and 3 months after CD5 CAR T cell infusion
  Objective response rate (ORR) is the percentage of subjects who have achieved CR, CRi or PR based on the National Comprehensive Cancer Network (NCCN) Guidelines Version 3.2023 of Acute Lymphoblastic Leukemia.
Phase 2- The incidence and severity of AEs | Up to 2 years
  The number of patients experiencing adverse events (AEs) and the severity of AEs will be evaluated.
Phase 2- Progression free survival (PFS) | Up to 2 years
  Progression-free survival (PFS) is defined as the time from the initial CD5 CAR T cell infusion to the date of progression or death for any cause.
Phase 2- Overall survival (OS). | Up to 2 years
  Overall survival (OS) is defined the time from the initial CD5 CAR T cell infusion to death for any cause.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Liquan Hospital, Shanghai, Shanghai Municipality
  - The General Hospital of Western Theater Command PLA, Chengdu, Sichuan